CLINICAL TRIAL: NCT00005995
Title: AE-941 (NEOVASTAT) Versus Placebo in Metastatic Renal Cell Carcinoma Patients Who Are Refractory to Immunotherapy
Brief Title: AE-941 in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000067999; AETERNA-AE-RC-99-02; CAN-CCI-ETH-00-32-17; CCF-IRB-3664; JGH-00023; UCMC-0006305; UPCC-2800
Record Dates: First submitted 2000-07-05; First posted 2004-02-12 (Estimated); Last update posted 2013-03-05 (Estimated); Status verified 2008-02

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — shark cartilage extract

INTERVENTIONS:
Drug: shark cartilage extract AE-941

SUMMARY:
RATIONALE: AE-941 may stop the growth of kidney cancer by stopping blood flow to the tumor.

PURPOSE: Randomized phase III trial to determine the effectiveness of AE-941 in treating patients who have metastatic kidney cancer that has not responded to biological therapy.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare survival of patients with metastatic renal cell carcinoma refractory to immunotherapy treated with AE-941 (Neovastat) versus placebo. II. Compare the time to progression and one-year survival rate of patients treated with this regimen. III. Determine the safety of this regimen in these patients. IV. Compare the overall tumor response rate, duration of response, and quality of life of patients treated with this regimen.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to number of organs with metastases (1 vs more than 1) and ECOG performance status (0 vs 1). Patients are randomized to one of two treatment arms. Arm I: Patients receive oral AE-941 (Neovastat) twice a day. Arm II: Patients receive oral placebo twice a day. Treatment continues in the absence of unacceptable toxicity or disease progression. Quality of life is assessed on day 1 and then every 8 weeks thereafter. Patients are followed every 4 weeks until disease progression and then every 8 weeks thereafter.

PROJECTED ACCRUAL: A total of 280 patients will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed renal cell adenocarcinoma Disease progression within 16 weeks after first-line therapy, which included interleukin-2 and/or interferon Metastatic disease not amenable to surgery Measurable and/or evaluable disease No more than one line of prior anticancer treatment for renal cell carcinoma No pure papillary cell tumor, mixed tumor containing predominantly sarcomatoid cells, Bellini carcinoma, medullary carcinoma, or chromophobe oncocytic tumor No brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: More than 3 months Hematopoietic: Platelet count at least 100,000/mm3 WBC at least 2,500/mm3 Hemoglobin at least 8 g/dL (epoetin alfa allowed) Hepatic: Not specified Renal: Calcium no greater than the upper limit of normal (ULN) (bisphosphonates allowed) Creatinine no greater than 2 times ULN Other: No other prior malignancy within past 5 years except basal cell carcinoma of the skin or carcinoma in situ of the cervix No severe allergy to fish or seafood No medical condition that would interfere with intake and/or absorption of study medication (e.g., gastrectomy or major intestinal resection) No significant medical or psychiatric condition that would preclude study Not pregnant Negative pregnancy test Fertile patients must use adequate contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics At least 1 month but no longer than 8 months since prior immunotherapy Chemotherapy: Not specified Endocrine therapy: At least 1 week since prior systemic corticosteroids for symptomatic treatment of renal cell carcinoma At least 28 days since prior medroxyprogesterone acetate No concurrent medroxyprogesterone acetate Concurrent corticosteroids for symptomatic treatment of neurological complications caused by renal cancer allowed Radiotherapy: Concurrent radiotherapy to symptomatic lesions for symptom relief allowed Surgery: See Disease Characteristics Concurrent surgical removal of symptomatic lesions for symptom relief allowed Other: At least 28 days since other prior experimental therapeutic agents At least 28 days since other prior shark cartilage products No other concurrent therapies for metastatic renal cell carcinoma No other concurrent shark cartilage products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-10; Primary Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Aeterna Zentaris, Québec, Quebec, Canada

REFERENCES:
- [Result] Escudier B, Choueiri TK, Oudard S, Szczylik C, Negrier S, Ravaud A, Chevreau C, Venner P, Champagne P, Croteau D, Dupont E, Hariton C, Bukowski RM. Prognostic factors of metastatic renal cell carcinoma after failure of immunotherapy: new paradigm from a large phase III trial with shark cartilage extract AE 941. J Urol. 2007 Nov;178(5):1901-5. doi: 10.1016/j.juro.2007.07.035. Epub 2007 Sep 17. PMID 17868728